CLINICAL TRIAL: NCT04511897
Title: Efficacy and Safety of An'Ningpai Enteric Soft Capsuleson in Stable Non-CF Bronchiectasis With Hypersecretion: a Open-label Randomized Controlled Trial
Brief Title: Efficacy and Safety of An'Ningpai Expectorant in Non-CF Bronchiectasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Chief of Department of Pulmonary and Critical Care Medicine, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200420
Record Dates: First submitted 2020-04-25; First posted 2020-08-13 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Bronchiectasis Adult
Keywords: Brochiectasis Adult; Hypersecretion; Exacerbation
MeSH Terms: interventions — Expectorants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): oral An'ningpai Enteric Soft Capsules (300 mg,three times daily) for 12 months.
  Interventions: Drug: An'ningpai
- Control group (No Intervention): No experimental durgs used.

INTERVENTIONS:
Drug: An'ningpai — An'ningpai Enteric Soft Capsules was a kind of expectorant, comprised with Eucalyptol, Limonene and Pinene. 300 mg, oral, three times daily for 12 months.
  Other Names: Expectorant
  Arms: Experimental group

SUMMARY:
The objective of this study was to assess whether the long-term use of oral An'Ningpai Enteric Soft Capsuleson (300 mg, three times daily, 12 months) might reduce the incidence of exacerbations and improve the quality of life in patients with Non-CF bronchiectasis.

DETAILED DESCRIPTION:
Mucus hypersecretion plays an essential role in bronchiectasis. It has been deduced that reducing the production of mucus or improving the clearance of sputum in the airway is the key to break down this "vicious cycle" and enhance the therapeutic efficacy for bronchiectasis.

The investgators aimed to assess whether the long-term use of oral An'Ningpai Enteric Soft Capsules (300 mg, three times daily) might reduce the rate of exacerbations and improve the quality of life in patients with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

1) subjects older than 18 ; 2)a diagnosis of bronchiectasis was according to the 2010 British Thoracic Society guidelines; 3) with hypersecretion ：high viscous sputum symptoms (sputum traits score 2-3 points) ;4) patients had least two exacerbations in the past year and were in a state for at least 4 weeks prior to randomization

Exclusion Criteria:

1) cystic fibrosis or other etiologies (such as immunodeficiency, allergic bronchopulmonary aspergillosis, traction bronchiectasis caused by emphysema, advanced pulmonary fibrosis, etc.); 2)primary diagnosis of COPD or asthma; 3)a history of severe cardiovascular disease; 4)comorbidity with liver disease, kidney disease, malignant tumor, gastric ulcer, or intestinal malabsorption; 5)a known allergy to Eucalyptol , Limonene and Pinene Enteric Soft Capsules; 6)pregnancy or lactation (for women);7)a history of prior macrolide use of more than 1 week; 8)and poor compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Numbers of acute exacerbation | one year

SECONDARY OUTCOMES:
The time to first exacerbation | one year
The volume of 24h sputum | Six months
Leicester Cough Questionnaire | Six months
  Cough Questionnaire for the degree of cough. The minimum value is 1 and maximum value is 21. Higher scores mean a better outcome
Questionnaire of life-Bronchiectasis | Six months
  Questionnaire for the life of bronchiectasis. The minimum value is 0 and maximum value is 100; higher scores indicate better health-related quality of life.
Incidence of diarrhea | Six months
  One of common adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jin-fu Xu, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China